CLINICAL TRIAL: NCT04270084
Title: Metabolic Optimization Through Diet/Lifestyle Improvements For Youth (MODIFY)
Brief Title: Metabolic Optimization Through Diet/Lifestyle Improvements For Youth
Acronym: MODIFY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's National Research Institute (Other)
Collaborators: University of California, Davis (Other); NutritionQuest (Unknown)
Responsible Party: Principal Investigator, Michele Mietus-Snyder, Associate Professor, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010790
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemias; Obesity
Keywords: cardiometabolic risk factors; lifestyle modification; visceral adiposity
MeSH Terms: conditions — Dyslipidemias; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Participants will be asked use a mobile health (m-health) app for 2 months. The app is designed to provide weekly education and motivation about healthful diet and physical activity behaviors in adolescents and their parent/adult caretaker. Both adolescent and parent/adult caretaker participants will use the app to enter weekly self-report data, set healthy eating and exercise goals, and receive educational and motivational content. Participants will conduct a weekly self-assessment of waist circumference, diet, and physical activity during the 2 month trial.
  Interventions: Behavioral: Alive-Family

INTERVENTIONS:
Behavioral: Alive-Family — All participants receive lifestyle modification through use of m-health app

SUMMARY:
The overarching goal of this study is to evaluate plasma ceramides (Cers) as early nutrition-sensitive biomarkers of metabolic health. The investigators will implement a diet and lifestyle intervention to improve cardiometabolic risk factors and test the corresponding change in Cer levels. The intervention will incorporate: a) family-level engagement, enrolling both adolescents and one parent/adult caretaker (PAC); and b) a behavior change mobile health (m-health) app, which will offer real-time support, education and monitoring of diet and activity.

DETAILED DESCRIPTION:
Dysregulated sphingolipid ceramide (Cer) metabolism impairs mitochondrial function, insulin sensitivity and vascular reactivity and has been identified as a central common pathway towards the dyslipidemia, central adiposity, hyperglycemia, and hypertension that define metabolic syndrome, characterized as cardiometabolic risk (CMR). The decrease in insulin sensitivity that occurs with age and predisposes to metabolic syndrome is preventable, a reflection of changes in body composition rather than the aging process itself. Ectopic fat, not fat mass per se, drives CMR, but despite mounting concern about rising prevalence of pediatric CMR in America and globally, the use of plasma Cer as potentially mechanistic biomarkers of ectopic fat and lipotoxicity has not been well explored. This may be driven in part by our incomplete understanding of i) the consequences of Cer dysregulation in pediatric CMR; ii) putative interactions between Cer and ectopic lipotoxicity; and iii) how lifestyle, notably nutrition, impacts Cer metabolism. Information in these areas may support use of plasma Cers as sensitive, prognostic biomarkers to guide more effective preventive lifestyle management of aberrant weight gain and associated CMR.

In preliminary work, the investigators compared plasma sphingolipid profiles in obese adolescents and their parent/adult caretakers (PAC). Data from this study demonstrated that Cers (notably C:14 and C:16) are associated with dyslipidemia in both adults and youth. The investigators also found that 2-mo of a daily nutrient bar supplementation (coupled with weekly group counseling and exercise) significantly decreased plasma Cers more effectively than counseling and physical exercise alone, without change in traditional biomarkers but the extent of Cer reduction correlated with improved dyslipidemia. The investigators also found that 10 days of dietary fructose reduction in obese pre-adolescents significantly lowers cers in direct proportion to the clearance of ectopic hepatic adiposity.

If study hypotheses are supported, these findings will identify sensitive Cer biomarkers of CMR with putative mechanistic insight to mitochondrial function requisite for insulin sensitivity, metabolic flexibility, lipolysis, and weight loss, that might therefore be used to monitor early success in lifestyle change trials.

ELIGIBILITY:
Adolescent inclusion criteria:

Aged 10 years to 18 years Dyslipidemia (TG/HDL-c >2.5 in non-Black males and >2.0 in females and Black males) Central adiposity (waist to height ratio > 0.5) Willingness to participate

Adult inclusion criteria:

Parent or adult caregiver of adolescent patient Central adiposity (waist to height ratio >0.5) Willingness to participate

Exclusion criteria (adolescent and parent) include

* Diabetes, genetic syndrome, stage II hypertension (systolic or diastolic BP > 95th percentile for age, sex, and height percentile + 12mm Hg or > 140/90, whichever is lower for subjects < 13 yr of age, > 140/90 for all > 13 yr of age, including PAC; history of hypertension controlled on stable medication regimen accepted)
* Medication use known to affect insulin sensitivity or lipid profiles, including metformin, statins, fibric acids or second generation atypical anti-psychotics (stable doses of stimulant or antidepressant therapy accepted)
* Current participation and unwillingness to cease activities related to a diet/exercise lifestyle modification program other than this program
* Any medical condition or syndrome with neurocognitive delay that would preclude active participation with the mobile health app
* Pregnancy or intention to become pregnant (as this will alter weight distribution)
* Inability to participate in moderate physical activity

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma ceramides | Change from Baseline level of plasma ceramides at 2 months
  S1P, C:14, and C:16

SECONDARY OUTCOMES:
Change in plasma lipids | Change from Baseline level at 2 months
  Plasma triglycerides, HDL-c, LDL-c
Change in plasma glucose | Change from Baseline level at 2 months
Change in plasma insulin | Change from Baseline level at 2 months
Change in plasma C-reactive protein (CRP) | Change from Baseline level at 2 months
Change in waist circumference | Change from Baseline level at 2 months
Change in BMI | Change from Baseline level at 2 months
  weight for height (Kg/M^2)
Change in physical activity | Change from Baseline level at 2 months
  Physical activity is assessed by self-report questionnaire. The activity questionnaire asks about frequency and duration of performance of a list of activities.
Change in diet | Change from Baseline level at 2 months
  Diet assessment by food frequency questionnaire (FFQ) to determine quantity and quality of macronutrients (carbs, protein, fat) and food groups (i.e. sugar sweetened beverages, fruits, vegetables, etc.) indexed as healthy eating score (Alternative Healthy Eating Index) on a scale of 2.5 to 87.5 with a higher score reflecting a more healthful diet.

OTHER OUTCOMES:
Mental health | Change from Baseline level at 2 months
  Mood and outlook will be assessed by self-report questionnaire: Patient Health Questionnaire for somatic symptoms, anxiety, and depression (PHQ-SADS) a continuous scale (0-86) with higher scores reflecting poorer mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mietus-Snyder, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No